CLINICAL TRIAL: NCT00149552
Title: Zinc Therapy in Zinc Deficient HIV Positive Drug Users
Brief Title: Zinc Therapy in HIV Infected Individuals Who Abuse Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marianna Baum, Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-14966-1; R01DA014966 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infections; Substance-Related Disorders
Keywords: Treatment Naive; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc gluconate (Active Comparator): Zinc supplementation
  Interventions: Dietary Supplement: zinc
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: zinc

INTERVENTIONS:
Dietary Supplement: zinc — supplementation with zinc gluconate

SUMMARY:
Zinc deficiency is prevalent in HIV infected individuals who abuse drugs. The purpose of this study is to determine if zinc therapy will prevent immune failure in HIV infected individuals who abuse drugs and have low plasma zinc levels.

DETAILED DESCRIPTION:
Low levels of zinc are associated with an increased risk of HIV-related death and opportunistic infections in HIV infected individuals. Drug users are especially susceptible to zinc deficiency. The purpose of this trial is to evaluate the effectiveness of zinc therapy in preventing immune failure in HIV infected individuals who abuse drugs.

This trial will last 30 months. Participants will be randomly assigned to receive either zinc supplements or placebo. Male participants will receive 15 mg of zinc and female participants will receive 12 mg of zinc. Clinical and laboratory study visits will occur at 3 or 6 month intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Drug User
* Blood zinc level greater than 0.35 mcg/mL and less than 0.75mcg/ml

Exclusion Criteria:

* Currently participating in an another clinical trial
* Blood selenium level less than 85 mcg/L
* Pregnant or intends to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2001-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Immune failure | For at least 6 months
  CD4 cell count <200 cells/uL

SECONDARY OUTCOMES:
Morbidity | For at least 6 months
  AIDS related morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Marianna K. Baum, PhD, Principal Investigator — Florida International University
Locations (1):
- Camillus House, Miami, Florida, United States

REFERENCES:
- [Derived] Baum MK, Lai S, Sales S, Page JB, Campa A. Randomized, controlled clinical trial of zinc supplementation to prevent immunological failure in HIV-infected adults. Clin Infect Dis. 2010 Jun 15;50(12):1653-60. doi: 10.1086/652864. PMID 20455705